CLINICAL TRIAL: NCT05587114
Title: A Retrospective Study to Compare Biomarker Expression of Exosomes Derived From Peripheral Blood and Primary Lung Cancer Drainage Pulmonary Blood in Lung Cancer Patients
Brief Title: Comparision of Various Biomarkers Between Peripheral and Pulmonary Blood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, Professor, Korea University Guro Hospital
Other Study IDs: 2020GR0340
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Diagnosis
Keywords: Exosome; biomarker; lung cancer; diagnosis; prognosis; liquid biopsy
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: frozen blood plasma samples — Analysis of various biomarkers using frozen blood samples

SUMMARY:
Lung cancer is a leading cause of cancer death worldwide. Early diagnosis is linked to a better prognosis. Further, surgical resection at the early stages of non-small cell lung cancer (NSCLC) results in markedly improved survival rates. Computed tomography (CT)- or bronchoscopy-guided needle biopsies are standard definitive diagnostic procedures for lung cancer and are used to obtain tissue for pathological examination. However, these procedures are invasive, difficult to repeat, expensive, and risk exposure to radiation. Conversely, liquid biopsies, such as circulating tumor cells (CTCs), circulating tumor DNA (ctDNA), and extracellular vesicles (EVs), are simple and less invasive procedures that can be repeated more frequently than tissue biopsies.

This study is a retrospective blood sample obtained and prospectively comparative analysis of various biomarkers (cancer markers, and exosome markers) derived from peripheral blood and pulmonary venous blood from patients who underwent lung cancer surgery.

And treatment monitoring using biomarkers compare with peripheral and pulmonary blood.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Korean nationality
* Patients who did not receive neoadjuvant therapy before surgery
* Patients not diagnosed with any other cancer before surgery
* Patients who agreed to the consent form for a donation of human materials during surgery

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, Koreans, regardless of gender, were studied for adults over 40 years of age.
  Blood plasma samples are optained from stored in the biobank of Korea University Guro Hospital or the Department of Thoracic and Cardiovascular Surgery of Korea University Guro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-13 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparative analysis of cancer marker concentrations in a peripheral vein and primary lung cancer outflow pulmonary vein | 2020 ~ 2025
  1. Comparative analysis of CEA and lung cancer-specific exosome marker concentrations in peripheral blood and pulmonary blood using ELISA assay
  2. Characterization of exosomes using western blot, NTA, and TEM analysis
Diagnostic analysis of lung cancer-specific exosome marker concentrations in a peripheral vein and primary lung cancer outflow pulmonary vein | 2020 ~ 2025
  1) Evaluation of the clinical usefulness of lung cancer diagnosis using lung cancer-specific exosome markers in peripheral vein blood and primary lung cancer outflow pulmonary vein-derived blood.

SECONDARY OUTCOMES:
Evaluation of lung cancer treatment monitoring using lung cancer-specific exosome biomarkers | 2020 ~ 2025
  Clinical evaluation of recurrence or cancer metastasis after treatment in patients who underwent lung cancer surgery using lung cancer-specific exosome biomarkers according to blood sample location (peripheral vein blood and primary lung cancer outflow pulmonary vein derived blood)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Koo Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No